CLINICAL TRIAL: NCT04190498
Title: Evaluation of the Prevalence of Sleep Apnea Syndrome in Patients With Hepatocellular Carcinoma
Brief Title: Sleep Apnoea Syndrome and Hepatocellular Carcinoma
Acronym: ECHAPS
Status: Withdrawn | Type: Observational
Why Stopped: the possibility of obtaining histological data is too low due to the lack of availability of biological samples
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.410; 2018-A02400-55 (Other: ID RCB)
Record Dates: First submitted 2019-11-04; First posted 2019-12-09 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Sleep Apnea, Obstructive; Hepatocellular Carcinoma; Non Alcoholic Steato Hepatitis
Keywords: Sleep Apnea, Obstructive; Hepatocellular carcinoma; Non Alcoholic Steato Hepatitis; hepatitis C virus
MeSH Terms: conditions — Sleep Apnea, Obstructive; Carcinoma, Hepatocellular; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NASH-related HCC: The study is focused on patients suffering from NASH-induced HCC. Each patient with NASH-related HCC will be paired with 2 patients with non NASH-related HCC (HCV-induced CHC).
  Interventions: Diagnostic Test: Nocturnal oximetry
- HCV-related HCC: HCV-related HCC has been chosen as control population for several reasons: HCV represent a common etiology of HCC; with a distinct pathophysiology distinct from that of post-NASH HCC; populations with post-NASH and post-HCV CHC share similar epidemiological characteristics.
  Interventions: Diagnostic Test: Nocturnal oximetry

INTERVENTIONS:
Diagnostic Test: Nocturnal oximetry — Diagnosis of OSA will be based on the 3% Oxygen Desaturation Index (IDO) obtained by home nocturnal oximetry. The oximetry recordings will be centralized in sleep laboratory of the University Hospital of Grenoble Alpes. Oximetry data will be analyzed by a technician from the sleep laboratory of the University Hospital of Grenoble Alpes

SUMMARY:
Obstructive sleep apnea (OSA), one of the most frequent respiratory diseases, could represent a major worsening factor in a non alcoholic steatohepatitis and neoplastic context. Our hypothesis is that OSA promotes the prevalence of HCC related to NASH. This national, multicenter study aims to compare the prevalence of OSA in a group of patient curatively resected for NASH-related HCC with a group of HCV-related HCC.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a common respiratory disease characterized by the occurrence of recurrent episodes of partial or total obstruction of the upper airway called hypopneas and apneas respectively. These episodes are associated with the repetitive occurrence of the desaturation-reoxygenation sequences, the so-called chronic intermittent hypoxia (IH) which is the major stimulus underlying main cardiovascular, metabolic consequences and pro-inflammatory state found in patients with OSA. Recent data from cohort studies have established that OSA is an even greater risk factor for cancer-related mortality. Hepatocellular carcinoma (HCC) is the second cancer related death worldwide and has an increasing impact in developed countries. The epidemic of metabolic syndrome (MS) plays a growing role in the occurrence of metabolic steatohepatitis (NASH) related HCC. Concerning transition from NASH to NASH-related HCC, neither the frequency nor the underlying mechanism are known. Very recently, a link between OSA (IH) and NASH has been highlighted. OSA and intermittent hypoxia should be a major worsening factor in a neoplastic context. Our hypothesis is that OSA promotes the prevalence of HCC in a context of NASH.

The objective is to compare the prevalence of OSA between patients with NASH-related and hepatitis C virus (HCV)-related HCC. In this type 3, cross-sectional, multicenter, national, non-randomized study patients suffering from a NASH-related or HCV-related hepatocellular carcinoma will be recruited. Investigators expect to show a higher prevalence of OSA in patients with HCC NASH-related but also a shorter overall survival. Complementary ex vivo studies on tumor samples will be conducted in order to explore the mechanisms by which OSA and IH would promote carcinogenesis

ELIGIBILITY:
Inclusion Criteria:

* Man and woman
* >18 years
* Diagnosis of NASH-induced HCC or HCV-induced HCC
* Patients treated by surgical excision
* Patients not opposed to the study

Exclusion Criteria:

* Patient refusal
* Alcohol consumption> 20g / day for women and> 30g / day for men
* Patient with HCV genotype 3
* Tumor vascular invasion identified preoperatively
* Other etiologies of hepatopathies (alcoholic, viral B, autoimmune, hemochromatosis)
* Other chronic respiratory diseases: chronic obstructive pulmonary disease, respiratory insufficiency
* Patient weight variation >5% since surgical treatment of his HCC
* Subject deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will prospectively included in the French Liver Biobanks network - INCa, BB-0033-00085 (CRB-Foie). Patients suffering from a NASH-related or HCV-related hepatocellular carcinoma who were only treated by surgery will be selected.
  Each NASH-related HCC patient will be adjusted with two HCV-related HCC patients based on a propensity score according to their age range, sex, BMI, tumor stage.
  For each patient, the duration of the study will be 1 month maximum, with only one visit for inclusion. Survival data at 12 and 24 months will be from the medical record and will not require a visit. The total duration of study will be 48 months.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
The study will compare OSA prevalence in a group of patient curatively resected for NASH-related HCC with a group of HCV-related HCC. | 2 years
  Number of patient presenting an obstructive apnea syndrome diagnosed by oxymetry

SECONDARY OUTCOMES:
The study will compare the 3% oxygen desaturation index between groups. | 2 years
  3% IDO represents the number of oxygen desaturation of at least 3% per hour of oxymetry recording, measured by one oximetry measurement during a single night at the patient's home.
The study will compare the 2% oxygen desaturation index between groups. | 2 years
  2% IDO represents the number of oxygen desaturation of at least 2% per hour of oxymetry recording, measured by one oximetry measurement during a single night at the patient's home.
The study will compare the 4% oxygen desaturation index between groups. | 2 years
  4% IDO represents the number of oxygen desaturation of at least 4% per hour of oxymetry recording, measured by one oximetry measurement during a single night at the patient's home.
This study will compare the number of micro-arousals between groups. | 2 years
  Micro-arousals associated with desaturation will be measured to characterize sleep fragmentation
This study will compare the time spent with a saturation less than 90 % between groups. | 2 years
  The time spent with a saturation less than 90 % (Tsat90 in second) to characterize oxygen desaturations and OSA severity
This study will compare the Pittsburgh Sleep Quality Index (PSQI) between groups. | 2 years
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality. Consisting of 19 items, the PSQI measures several different aspects of sleep. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
This study will compare the Epworth Sleepiness Score between groups. | 2 years
  The Epworth sleepiness scale (ESS) is a self-administered questionnaire that's routinely used by doctors to assess daytime sleepiness. The person filling in the questionnaire rates how likely they are to doze off during the day in 8 different situations.The test evaluate the tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing.
The study will compare the prevalence of OSA in patients with NASH-induced CHC with cirrhotic context compared to NASH-induced CHC patients without cirrhosis. | 2 years
  Number of patient presenting an obstructive apnea syndrome diagnosed by oxymetry in both subpopulations: cirrhotic and non-cirrhotic.
The study will compare the NAFLD Activity Score (NAS score) between OSA and non-OSA subgroups of NASH patients. | 2 years
  NAFLD Activity Score includes the degree of steatosis, hepatocyte ballooning, lobular inflammation and fibrosis. Nas score is between 0 and 16.
The study will compare the Brunt score between OSA and non-OSA subgroups of NASH patients. | 2 Years
  The Brunt score for NASH patients is used to evaluate fibrosis stage. The score is between 1 and 4.
The study will compare the METAVIR score data between HCV OSA and HCV non-OSA patients. | 2 Years
  The METAVIR score is used to evaluate fibrosis stage for HCV patients. The score is between 0 and 4.
The study will compare BCLC classification of HCC tumor between groups. | 2 years
  Tumor stage evaluated by BCLC classification scale :0,A,B,C and D values (0 for Stage 0 Very early stage, D for terminal stage)
The study will compare HCC tumor size between each groups. | 2 years
  Tumor size (expressed in cm) is asociated to HCC prognostic the size of the tumor is associated with the prognosis of the HCC
The study will compare HCC tumor differentiation degree between groups. | 2 years
  The tumor differentiation is classified in 3 levels: low, moderate or high level of tumor differentiation
The study will compare vascular invasion of HCC tumor between groups. | 2 years
  Presence or absence of tumor vascular invasion
The study will compare the number of satellite nodules of HCC between between groups. | 2 years
  Number of tumoral satellite nodules (multifocality)
The study will compare plasma alpha fetoprotein level between groups. | 2 years
  Plasma alpha fetoprotein (AFP) level expressed in ng/ml
The study will compare overall survival rate between groups. | 2 years
  Overall survival at 1 and 2 years will be collected.
The study will compare tumor-free survival rate between groups. | 2 years
  Tumor-free survival at 1 and 2 years will be collected.
The study will compare non-recurrence-free survival rate between groups. | 2 years
  Non-recurrence-free survival at 1 and 2 years will be retrospectively or prospectively collected.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, MD,PHD, Principal Investigator — University Hospital, Grenoble; Thomas Decaens, MD,PHD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Minovés-Kotzki, La Tronche, Rhones-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided